CLINICAL TRIAL: NCT03138330
Title: Validation of Dietary Patterns and Inflammatory Salivary Biomarkers Among Healthy Toddlers of 15-36 Months Old in Singapore
Brief Title: Validation of a Food Frequency Questionnaire
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SGP. 1.A/A/3, PIEC2015/023.
Record Dates: First submitted 2017-02-13; First posted 2017-05-03 (Actual); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: this study is observational, it is not an intervention

SUMMARY:
The purpose of this study is to collect nutritional information from young children aged 15-36 months to validate a newly developed food frequency questionnaire.

DETAILED DESCRIPTION:
The primary purpose of this study is to validate a semi-quantitative food frequency questionnaire (FFQ) against a reference method (2-day weighed food records) in a sample of young children aged 15-36 months.

In addition to dietary data, the investigators also collected information on parental demographics, toddler health with regards to allergies and intolerance, parental feeding practices, parent and child weight and height and lastly, saliva samples to study inflammatory markers.

Therefore, in addition to the validation of the FFQ- the data will also be used to study associations between dietary patterns, food and nutrient intake and (i) parental feeding practices and (ii) inflammatory biomarkers from saliva

ELIGIBILITY:
Inclusion Criteria:

1. 15-36 months old boys and girls who are healthy
2. Toddlers who are from either Chinese, Malay or Indian ethnic group

Exclusion Criteria:

1. Toddlers with any acute or chronic illness, such as chronic inflammatory bowel disease, or illness that negatively affects food intake (e.g. Crohn's disease or ulcerative colitis).
2. Toddlers with history of antibiotics used in the last 1 week before the study.
3. Toddlers with history of vaccination in the last 2 weeks before the study
4. Toddlers with one or both parents of Caucasian origin.

Ages: 15 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who are aged 15-36 months and of Chinese, Indian or Malay ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sandalova, PhD, Principal Investigator — Danone Nutricia Early Life Nutrition; Smita Nambiar-Mann, PhD, Study Chair — Danone Nutricia Early Life Nutrition

IPD SHARING:
Plan to Share IPD: Undecided
the whole data set (without traceability to the participant) may be available for other researchers for secondary analyses

REFERENCES:
- [Derived] Allan C, Abdul Kader UH, Ang JYY, Muhardi L, Nambiar S. Relative validity of a semi-quantitative food frequency questionnaire for Singaporean toddlers aged 15-36 months. BMC Nutr. 2018 Dec 11;4:42. doi: 10.1186/s40795-018-0252-9. eCollection 2018. PMID 32153903

RESULTS

PARTICIPANT FLOW:
Groups:
- FFQ Group: Ninety-one parents of Singaporean toddlers completed the sqFFQ and a 2-day weighed food record as the reference method.
Period: Overall Study
Arm/Group | FFQ Group
Started | 95
Completed | 91
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- FFQ Group: The study included toddlers of 15-39 months of age of Chinese, Malay, or Indian ethnicity in Singapore.
Arm/Group | FFQ Group
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 23 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 44
Region of Enrollment [Number; unit: participants]
  Singapore | 91

OUTCOME MEASURES:

1. Primary Outcome: Validated Food Frequency Questionnaire
Description: Ninety-one parents completed the sqFFQ and a 2-day weighed food record as the reference method. Intake of energy and nutrients (energy, carbohydrates, fat, protein, fibre, sugars, calcium and iron) were determined for each method and compared using Pearson correlations.
Time Frame: up to 1 month
Population: Ninety-one parents of Singaporean toddlers who completed the sqFFQ and a 2-day weighed food record. Here pearson correlation between the two methods (FFQ and food diary) is presented.
Measure: Number; unit: Pearson correlation
Arm/Group | FFQ Group
Number analyzed (Participants) | 91
Pearson correlation
  total Energy | 0.39
  Protein | 0.35
  total fat | 0.28
  total carbohydrates | 0.32
  sugars | 0.42
  fibre | 0.56
  Calcium | 0.62
  Iron | 0.28

2. Secondary Outcome: Salivary Inflammatory Biomarkers
Description: C-reactive protein, salivary IgA, alpha amylase
Time Frame: up to 1 month
Population: Subjects who had sufficient saliva sample for analysis. There was not sufficient saliva sample to measure the CRP values, thus CRP values are not reported.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | FFQ Group
Number analyzed (Participants) | 76
ug/ml
  IgA | 119314 (157368)
  Amylase | 79 (60)

ADVERSE EVENTS:
Arm/Group | FFQ Group
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes